CLINICAL TRIAL: NCT07026084
Title: Effects of Biofeedback-Guided Training on Muscle Strength and Postural Alignment in Upper Cross Syndrome.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Riphah IU Shizra Tayyab
Record Dates: First submitted 2025-06-11; First posted 2025-06-18 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Upper Extremity Problem; Muscle Weakness; Postural Kyphosis
Keywords: upper cross syndrome; forward head posture; young adults; bio feedback guided training; postural alignment
MeSH Terms: conditions — Muscle Weakness; Oculocerebral hypopigmentation syndrome type Preus

STUDY DESIGN:
Intervention Model Description: comparison based study on effects of bio feedback guided training and conventional exercise prorocol on muscle strength and postural training in upper cross syndrome
Who Masked: Participant, Investigator
Masking Description: Participants will be masked by using sealed envolpe method
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Biofeedback-Guided Strength Training:
  Hot Pack: Applied for 10 minutes, mild warmth sensation to relax muscles and prepare for exercise.
  1. BPU (Biofeedback Pressure Unit): performed at 5 pressure levels (22, 24, 26, 28, 30 mmHg).
  Each level involves a 10-second hold, with 30 seconds rest between levels.
  Targeted muscles:
  * Deep Cervical Flexors (Capitus Longus, Capitus Colli).
  * Rhomboids
  * Trapezius Total duration (BPU): 20 minutes/session, performed 3 times/week.
  Interventions: Other: Bio feedback training
- Control Group (Active Comparator): Conventional Therapy:
  Hot Pack: Applied for 10 minutes, mild warmth sensation to relax muscles and prepare for exercise.
  EXERCISE PROGRAM:
  * 1. Supine: Neck curl with Chin Tucks (Deep Cervical Flexors Capitus Longus, Capitus Colli): 10 reps/session, holding each for 5 seconds.
  * 2. Sitting: Chin tuck with Head pushing against palm.
  * 3. Chin Up (Middle and Lower Trapezius): 10 reps/session, holding each for 5 seconds.
  * 4. Scapular Squeezes (Rhomboids): 2-3 sets of 10 reps/session, holding each for 5 seconds
  * 5. Doorway Pectoral Stretch (pect major) 2-3 reps, 30 sec hold (36) Total duration: 20 minutes/session, performed 3 times/week.
  Interventions: Other: conventional exercise program

INTERVENTIONS:
Other: Bio feedback training — Hot Pack: Applied for 10 minutes, mild warmth sensation to relax muscles and prepare for exercise.
  1. BPU (Biofeedback Pressure Unit): performed at 5 pressure levels (22, 24, 26, 28, 30 mmHg).
  Each level involves a 10-second hold, with 30 seconds rest between levels.
  Targeted muscles:
  * Deep Cervical Flexors (Capitus Longus, Capitus Colli).
  * Rhomboids
  * Trapezius Total duration (BPU): 20 minutes/session, performed 3 times/week.
  Arms: Experimental Group
Other: conventional exercise program — Hot Pack: Applied for 10 minutes, mild warmth sensation to relax muscles and prepare for exercise.
  EXERCISE PROGRAM:
  * 1. Supine: Neck curl with Chin Tucks (Deep Cervical Flexors Capitus Longus, Capitus Colli): 10 reps/session, holding each for 5 seconds.
  * 2. Sitting: Chin tuck with Head pushing against palm.
  * 3. Chin Up (Middle and Lower Trapezius): 10 reps/session, holding each for 5 seconds.
  * 4. Scapular Squeezes (Rhomboids): 2-3 sets of 10 reps/session, holding each for 5 seconds• 5. Doorway Pectoral Stretch (pect major) 2-3 reps, 30 sec hold (36)Total duration: 20 minutes/session, performed 3 times/week.
  Arms: Control Group

SUMMARY:
This randomized controlled trial investigates the effects of biofeedback-guided training versus conventional therapy on muscle strength and postural alignment in patients with Upper Cross Syndrome. The study includes adults aged 25-45 years meeting diagnostic criteria for UCS, such as weak deep cervical flexors, restricted cervical ROM, forward head posture, increased thoracic kyphosis, and chronic neck pain >3 months. Participants are divided into two groups: Group A biofeedback training and Group B conventional therapy, receiving 12 sessions over 4 weeks ,3sessions/week. Assessments are conducted at baseline, post-1st session, and weekly intervals using standardized measures.The study aims to compare the efficacy of biofeedback-guided training in improving strength and posture in UCS patients.

DETAILED DESCRIPTION:
Prolonged sitting and repetitive movements, common in desk jobs, poor ergonomics, and sedentary lifestyles, can lead to poor posture, discomfort, pain, and muscle or joint disability. A frequent result of poor posture is Upper Cross Syndrome, characterized by imbalances between upper body muscle groups. In Upper Cross Syndrome, overactive muscles like the pectoralis major, upper trapezius, and levator scapulae become tight, while the deep neck flexors, middle and lower trapezius, serratus anterior, and rhomboids weaken, disrupting movement patterns and increasing injury risk. Dr. Janda's 1988 model categorized muscles into postural (tonic) muscles, prone to tightness, and phasic muscles, prone to weakness. Upper cross Syndrome commonly causes neck, shoulder, and upper back pain, along with discomfort in the shoulder blades and neck stiffness.

Upper Cross Syndrome symptoms include neck, shoulder, and upper back pain, and can lead to forward head posture , increased thoracic kyphosis, and loss of cervical lordosis. Forward head posture, seen in 60% of individuals aged 20 to 50, causes neck strain, reduced mobility, and pain. With the rise of technology use, Upper cross syndrome has become more prevalent. Individuals often lean forward to view screens, exacerbating posture-related issues. Studies show Upper cross syndrome prevalence in IT professionals (67%), students (37.1%) and laundry workers (28%). Prevalence across different groups ranges from 11% to 60%. This condition leads to pain, discomfort, and reduced quality of life, prompting the need for effective treatment.

Effective manual therapy techniques for treating Upper Cross Syndrome aim to alleviate muscle tension, improve mobility, and correct postural imbalances. These include joint mobilization and manipulation, which restore normal motion and reduce pain, and soft tissue mobilization techniques like myofascial release and trigger point therapy that target tight muscles to enhance blood flow and reduce tension. Active Release Techniques identify and release muscle adhesions through specific movements and therapist-applied pressure, while transverse massage uses friction across muscle fibers to break down adhesions and promote healing. Post-Isometric Relaxation helps enhance flexibility and reduce tightness by contracting and stretching muscles, and neuro-mobilization addresses nerve entrapments commonly associated with Upper cross syndrome to alleviate pain.

A growing body of research has explored the effectiveness of various interventions for managing Upper cross syndrome, including manual therapy, and biofeedback-guided strength training. Karthi et al. found that motor control training of deep neck flexors using pressure biofeedback significantly reduced pain and disability, highlighting the efficacy of biofeedback in improving muscle activation and posture. Similarly, Ashfaq et al. demonstrated that cranio-cervical flexion training with biofeedback enhanced muscular endurance and reduced neck pain more effectively than conventional methods. These findings align with the clinical utility of biofeedback in correcting postural imbalances, a key feature of UCS. In addition, ART, which targets muscle adhesions and soft tissue dysfunction, has shown promise in improving range of motion and alleviating pain in UCS patients (Kang et al., 2016).Manual therapy techniques like joint mobilization and soft tissue manipulation are also effective in restoring normal movement patterns and reducing discomfort. Gumuscu et al. further supported these findings by showing that combining conventional program i.e. stabilization exercises with stretching and strengthening improved posture and respiratory function in office workers with forward head posture, suggesting that integrated approaches could enhance outcomes in Upper cross syndrome management.

Strength training has been widely used to correct Upper cross syndrome by targeting weak muscle groups, particularly DCFs. Studies have shown that resistance exercises can significantly improve posture and reduce associated pain by enhancing muscle endurance and correcting imbalances. However, conventional strength training lacks real-time feedback mechanisms, not providing neuromuscular control, potentially leading to compensatory movements and suboptimal outcomes.

ELIGIBILITY:
Inclusion Criteria:

* • Adults aged 25-45 years with both genders.

  * Individuals meeting the following diagnostic criteria for upper cross syndrome will be included:
  * Reduced strength of deep cervical flexors = unable to maintain pressure beyond 22-24 mm Hg (assessed via cranio-cervical flexion test).
  * Limited cervical range of motion (Flexion: < 80 degrees, Extension: < 70 degrees, Rotation: < 90 degrees on both sides, Lateral Flexion: < 20 degrees)
  * Postural deviations: forward head posture (CVA <50 degrees), increased thoracic kyphosis (via flexi curve >45 degrees).
  * Neck pain with a duration of over 3 months

Exclusion Criteria:

* • History of recent neck surgery or injury.

  * Patients with neurological disorders affecting muscle tone.
  * Involvement in other physical therapy programs focused on UCS.
  * Diagnosed musculoskeletal condition that could impact muscle performance.

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 56 (Estimated)
Dates: Start 2025-08-11 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
cranio-cervical flexion test | baseline to 4th week
  craniocervical flexion test to measure strength and endurance of Deep cervical flexors. it ranges from 20 mm of hg to 30 mm of Hg based on increased strength

SECONDARY OUTCOMES:
NPRS | total of 5 measurements taken at baseline, at the end of 1st, 2nd , 3rd and 4th week
  Pain is measured through NPRS scale. it has 11 level points from 0-10. where 0 indicate no pain and 10 indicate un-bearable pain
NECK DISABILITY INDEX | total of 5 measurements taken at baseline, at the end of 1st, 2nd , 3rd and 4th week
  neck disability is measured through NDI. it has score from 0-50. where 0 indicate low disability and 50 indicate total disability
cervical Flexion | baseline to 4th week
  A goniometer is a reliable and valid tool for assessing joint angles. cervical flexion is mesaured when the chin tries to touch the chest. it ranges from o-40 degrees.
cervical Extension | baseline to 4th week
  A goniometer is a reliable and valid tool for assessing joint angles. cervical extension is mesaured when the person tries to look up to the roof as max as he/she can go. it ranges from 0-70 degrees.
cervical Rt rotation | baseline to 4th week
  A goniometer is a reliable and valid tool for assessing joint angles. cervical Rt rotation is measured when the person face tries to look to the right
cervical Lt rotation | baseline to 4th week
  A goniometer is a reliable and valid tool for assessing joint angles. cervical Lt rotation is measured when the person face tries to look to the left. it ranges from 0-45 degrees
cervical Lt flexion | baseline to 4th week
  A goniometer is a reliable and valid tool for assessing joint angles. cervical Lt flexion is measured when the lt ear tries to touch to the shoulder
cervical Rt flexion | baseline to 4th week
  A goniometer is a reliable and valid tool for assessing joint angles. cervical Rt flexion is measured when the Rt ear tries to touch to the shoulder.

CONTACTS AND LOCATIONS:
Overall Officials: Aisha Razzaq, PHD*, Principal Investigator — Riphah International University
Locations (1):
- Watch Guard Tech, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No